CLINICAL TRIAL: NCT01048671
Title: Collection of Data on the Management of HIV-1 Patients Treated With Antiretroviral Combination Therapy Including the HIV Integrase Inhibitor Raltegravir
Brief Title: Management of Human Immunodeficiency Virus 1 (HIV-1) Participants Treated With Antiretroviral (ARV) Combination Therapy Including Raltegravir (MK-0518-138)
Acronym: RACING
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 0518-138; MK0518-138
Record Dates: First submitted 2010-01-12; First posted 2010-01-14 (Estimated); Results first posted 2014-02-14 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-10

CONDITIONS: HIV Infections
Keywords: HIV
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Antiretroviral combination therapy including raltegravir: Participants received ARV combination treatment including raltegravir. Treatment of participants was at the discretion of the investigator who provided standard care in a real life setting.
  Interventions: Drug: Raltegravir; Drug: ARV (non-raltegravir)

INTERVENTIONS:
Drug: Raltegravir — Raltegravir was administered in combination with ARV therapies at the discretion of the investigator in accordance with the product label. The recommended dose of raltegravir is 400 mg twice daily.
  Other Names: Isentress
Drug: ARV (non-raltegravir) — ARV treatments were administered in combination with raltegravir at the discretion of the investigator in accordance with the product labels, and could include nucleoside reverse-transcriptase inhibitor, non-nucleoside reverse-transcriptase inhibitor, protease inhibitor, entry inhibitor, and integrase inhibitor catagories.

SUMMARY:
To evaluate the management of HIV-1 participants treated with antiretroviral combination therapy including the integrase inhibitor raltegravir, all across the country of France.

ELIGIBILITY:
Inclusion Criteria:

* Participant Infected With HIV-1.
* Participant for whom raltegravir therapy has been decided and started less than 30 days prior to inclusion in the study.
* Participant who has received oral and written information about the study and who has agreed to the computer processing of his/her personal data.

Exclusion Criteria:

* Participant taking part in a clinical trial to assess raltegravir.
* Participant in whom raltegravir treatment was started more than 30 days ago.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participant Infected With HIV-1
Sampling Method: Non-Probability Sample
Enrollment: 482 (Actual)
Dates: Start 2010-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 482 participants included in the trial, 2 were excluded from analysis. A single treatment arm was specified in the study, but participants were sub grouped by their prior ARV experience at Baseline (ARV naïve, suppressed, or virological failure) for analysis.
Groups:
- ARV naïve at Baseline: ARV naïve participants had no previous experience with ARV. Participants received ARV combination treatment including raltegravir. Treatment of participants was at the discretion of the investigator who provided standard care in a real life setting.
- Suppressed at Baseline: Suppressed participants had previous ARV experience and had a viral load <50 ribonucleic acid (RNA) copies/mL at Baseline. Participants received ARV combination treatment including raltegravir. Treatment of participants was at the discretion of the investigator who provided standard care in a real life setting.
- Virological Failure at Baseline: Virological failure participants had previous ARV experience and had a viral load >50 RNA copies/mL at Baseline. Participants received ARV combination treatment including raltegravir. Treatment of participants was at the discretion of the investigator who provided standard care in a real life setting.
Period: Overall Study
Arm/Group | ARV naïve at Baseline | Suppressed at Baseline | Virological Failure at Baseline
Started | 66 | 264 | 152
Completed | 66 | 263 | 151
Not Completed | 0 | 1 | 1
Not completed — Protocol Violation | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Suppressed at Baseline: Suppressed participants had previous ARV experience and had a viral load <50 RNA copies/mL at Baseline. Participants received ARV combination treatment including raltegravir. Treatment of participants was at the discretion of the investigator who provided standard care in a real life setting. One participant in this subgroup was excluded from analysis because of protocol violation (inclusion criterion not met).
- Virological Failure at Baseline: Virological failure participants had previous ARV experience and had a viral load >50 RNA copies/mL at Baseline. Participants received ARV combination treatment including raltegravir. Treatment of participants was at the discretion of the investigator who provided standard care in a real life setting. One participant in this subgroup was excluded from analysis because of protocol violation (inclusion criterion not met).
- Total: Total of all reporting groups
Arm/Group | ARV naïve at Baseline | Suppressed at Baseline | Virological Failure at Baseline | Total
Number analyzed (Participants) | 66 | 263 | 151 | 480
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.9 (12.0) | 47.3 (10.1) | 46.5 (10.4) | 46.4 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 91 | 65 | 173
  Male | 49 | 172 | 86 | 307
Time Since Human Immunodeficiency Virus (HIV) Infection Diagnosis [Mean (Standard Deviation); unit: Years] | 2.8 (4.7) | 13.0 (7.0) | 11.6 (7.5) | 11.1 (7.7)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Receiving Antiretroviral Treatments Administered With Raltegravir
Description: Participants received ARV combination treatment including raltegravir. Treatment of participants was at the discretion of the investigator who provided standard care in a real life setting. ARV treatments included any nucleoside reverse transcriptase inhibitors (NRTIs), combination of tenovir/emitricitabine (FTC/TDF), combination of lamivudine/abacavir (3TC/ABC), protease inhibitors, and others.
Time Frame: Up to 25 months after start of raltegravir treatment
Population: Two participants were excluded for protocol violation (inclusion criterion not met) and data were missing for 3 additional participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Antiretroviral Combination Therapy Including Raltegravir
Number analyzed (Participants) | 477
Percentage of participants
  FTC/TDF + raltegravir | 44.4
  3TC/ABC + raltegravir | 14.0
  Other 2 NRTIs + raltegravir | 1.3
  Mulitple (>=3 ) ARV therapies + raltegravir | 15.7
  Protease inhibitor + raltegravir | 8.8
  Other strategies (each <5%) | 15.7

2. Primary Outcome: Percentage of Participants Responding to Treatment: All Treated Participants
Description: Response to treatment was defined as a viral load <50 RNA copies/mL
Time Frame: 24 months after start of raltegravir treatment
Population: All participants with a viral load assessment available at 24 months were included in the analysis. A single treatment arm was specified in the study, but participants were sub grouped by their prior ARV experience at Baseline (ARV naïve, suppressed, or virological failure) for analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Suppressed at Baseline: Suppressed participants had previous ARV experience and had a viral load <50 RNA copies/mL at Baseline. Participants received ARV combination treatment including raltegravir. Treatment of participants was at the discretion of the investigator who provided standard care in a real life setting.
- All Participants: Participants received ARV combination treatment including raltegravir. Treatment of participants was at the discretion of the investigator who provided standard care in a real life setting.
Arm/Group | ARV naïve at Baseline | Suppressed at Baseline | Virological Failure at Baseline | All Participants
Number analyzed (Participants) | 52 | 230 | 125 | 407
Percentage of participants | 94.2 [87.9 to 100.6] | 94.3 [91.4 to 97.3] | 71.2 [63.3 to 79.1] | 87.2 [84.0 to 90.5]

3. Primary Outcome: Percentage of Participants Responding to Treatment: Participants Still Receiving Raltegravir Treatment at Month 24
Description: Response to treatment was defined as a viral load <50 RNA copies/mL
Time Frame: 24 months after start of raltegravir treatment
Population: All participants with a viral load assessment available and receiving raltegravir treatment at 24 months were included in the analysis. A single treatment arm was specified in the study, but participants were sub grouped by their prior ARV experience at Baseline (ARV naïve, suppressed, or virological failure) for analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ARV naïve at Baseline | Suppressed at Baseline | Virological Failure at Baseline | All Participants
Number analyzed (Participants) | 39 | 194 | 94 | 327
Percentage of participants | 94.9 [87.9 to 101.8] | 95.4 [92.4 to 98.3] | 77.7 [69.2 to 86.1] | 90.2 [87.0 to 93.4]

4. Primary Outcome: Mean Change From Baseline in Cluster of Differentiation 4 (CD4) Cell Count: All Treated Participants
Time Frame: Baseline and 24 months after start of raltegravir treatment
Population: All participants with a CD4 cell count available at 24 months were included in the analysis. A single treatment arm was specified in the study, but participants were sub grouped by their prior ARV experience at Baseline (ARV naïve, suppressed, or virological failure) for analysis.
Measure: Mean (95% Confidence Interval); unit: cells/mm^3
Arm/Group | ARV naïve at Baseline | Suppressed at Baseline | Virological Failure at Baseline | All Participants
Number analyzed (Participants) | 55 | 229 | 123 | 407
cells/mm^3 | 260.58 [208.75 to 312.41] | 47.97 [19.57 to 76.36] | 149.98 [113.71 to 186.26] | 107.53 [85.80 to 129.29]

5. Primary Outcome: Mean Change From Baseline in CD4 Cell Count: Participants Still Receiving Raltegravir Treatment at Month 24
Time Frame: Baseline and 24 months after start of raltegravir treatment
Population: All participants with a CD4 cell count available and receiving raltegravir treatment at 24 months were included in the analysis. A single treatment arm was specified in the study, but participants were sub grouped by their prior ARV experience at Baseline (ARV naïve, suppressed, or virological failure) for analysis.
Measure: Mean (95% Confidence Interval); unit: cells/mm^3
Arm/Group | ARV naïve at Baseline | Suppressed at Baseline | Virological Failure at Baseline | All Participants
Number analyzed (Participants) | 39 | 194 | 91 | 324
cells/mm^3 | 285.05 [219.96 to 350.15] | 49.21 [16.38 to 82.03] | 150.87 [110.88 to 190.86] | 106.15 [80.87 to 131.43]

6. Secondary Outcome: Number of Participants With at Least One Adverse Event
Description: An adverse event was defined as any untoward, undesired, or unplanned clinical event in the form of physical signs, symptoms, disease, laboratory or physiological observations in a participant administered the sponsor's product whether or not related to the use of the product.
Time Frame: Up to 25 months after start of raltegravir treatment
Population: Participants enrolled and not excluded for a protocol violation were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Antiretroviral Combination Therapy Including Raltegravir
Number analyzed (Participants) | 480
Participants | 287

ADVERSE EVENTS:
Description: Two participants were excluded from the analysis because of protocol violation (inclusion criterion not met).
Arm/Group | Antiretroviral Combination Therapy Including Raltegravir
Serious Adverse Events (participants affected / at risk) | 66/480
Other Adverse Events (participants affected / at risk) | 27/480
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Antiretroviral Combination Therapy Including Raltegravir (N=480)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1)
FEBRILE BONE MARROW APLASIA (Blood and lymphatic system disorders) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1)
ANGINA PECTORIS (Cardiac disorders) | 1 (1)
CARDIAC DISORDER (Cardiac disorders) | 1 (1)
CARDIAC FAILURE (Cardiac disorders) | 1 (1)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 1 (1)
CARDIOGENIC SHOCK (Cardiac disorders) | 1 (1)
CORONARY ARTERY STENOSIS (Cardiac disorders) | 1 (1)
PERICARDIAL EFFUSION (Cardiac disorders) | 1 (1)
DEAFNESS (Ear and labyrinth disorders) | 1 (1)
ASCITES (Gastrointestinal disorders) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 1 (1)
DIARRHOEA HAEMORRHAGIC (Gastrointestinal disorders) | 1 (1)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1)
INGUINAL HERNIA (Gastrointestinal disorders) | 1 (1)
INGUINAL HERNIA STRANGULATED (Gastrointestinal disorders) | 1 (2)
NAUSEA (Gastrointestinal disorders) | 1 (1)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1)
ASTHENIA (General disorders) | 2 (2)
CHEST PAIN (General disorders) | 1 (1)
DEATH (General disorders) | 1 (1)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 2 (2)
INFLUENZA LIKE ILLNESS (General disorders) | 1 (1)
MULTI-ORGAN FAILURE (General disorders) | 1 (1)
OEDEMA PERIPHERAL (General disorders) | 1 (1)
PAIN (General disorders) | 1 (1)
SWELLING (General disorders) | 1 (1)
CHOLESTASIS (Hepatobiliary disorders) | 1 (1)
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 1 (2)
CRYOGLOBULINAEMIA (Immune system disorders) | 1 (1)
IMMUNE RECONSTITUTION SYNDROME (Immune system disorders) | 1 (1)
ABSCESS NECK (Infections and infestations) | 1 (1)
BRONCHOPNEUMONIA (Infections and infestations) | 1 (1)
CANDIDA SEPSIS (Infections and infestations) | 1 (1)
CEREBRAL TOXOPLASMOSIS (Infections and infestations) | 1 (1)
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 1 (1)
CYTOMEGALOVIRUS CHORIORETINITIS (Infections and infestations) | 1 (1)
HISTOPLASMOSIS (Infections and infestations) | 1 (2)
HISTOPLASMOSIS DISSEMINATED (Infections and infestations) | 1 (1)
LUNG INFECTION (Infections and infestations) | 1 (1)
MENINGITIS VIRAL (Infections and infestations) | 1 (1)
MYCOBACTERIAL INFECTION (Infections and infestations) | 1 (1)
PNEUMOCYSTIS JIROVECI PNEUMONIA (Infections and infestations) | 2 (2)
POST PROCEDURAL INFECTION (Infections and infestations) | 1 (1)
PULMONARY SEPSIS (Infections and infestations) | 1 (1)
PYELONEPHRITIS (Infections and infestations) | 1 (1)
SEPSIS (Infections and infestations) | 1 (1)
SEPTIC SHOCK (Infections and infestations) | 2 (2)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1 (1)
TOOTH INFECTION (Infections and infestations) | 1 (1)
ACCIDENT (Injury, poisoning and procedural complications) | 1 (1)
ALCOHOL POISONING (Injury, poisoning and procedural complications) | 1 (1)
DEVICE FAILURE (Injury, poisoning and procedural complications) | 1 (1)
FOOT FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
HEAD INJURY (Injury, poisoning and procedural complications) | 1 (1)
POST-TRAUMATIC PAIN (Injury, poisoning and procedural complications) | 1 (1)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 1 (1)
SCAN (Investigations) | 1 (1)
TRANSAMINASES INCREASED (Investigations) | 1 (1)
WEIGHT DECREASED (Investigations) | 1 (1)
CACHEXIA (Metabolism and nutrition disorders) | 1 (1)
MALNUTRITION (Metabolism and nutrition disorders) | 1 (2)
MITOCHONDRIAL CYTOPATHY (Metabolism and nutrition disorders) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1)
FISTULA (Musculoskeletal and connective tissue disorders) | 1 (1)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1 (1)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1)
OSTEOPENIA (Musculoskeletal and connective tissue disorders) | 1 (1)
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 1 (1)
CARCINOMA IN SITU (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
CERVIX CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
ENDOMETRIAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
NON-HODGKIN'S LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OROPHARYNGEAL CANCER STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 (2)
HEADACHE (Nervous system disorders) | 3 (4)
HEMIPARESIS (Nervous system disorders) | 1 (1)
ISCHAEMIC STROKE (Nervous system disorders) | 1 (1)
ANXIETY (Psychiatric disorders) | 1 (1)
DEPRESSION (Psychiatric disorders) | 5 (5)
LIBIDO DECREASED (Psychiatric disorders) | 1 (1)
NEGATIVE THOUGHTS (Psychiatric disorders) | 1 (1)
PARANOIA (Psychiatric disorders) | 1 (1)
SCHIZOPHRENIA (Psychiatric disorders) | 1 (1)
SUICIDE ATTEMPT (Psychiatric disorders) | 4 (4)
RENAL FAILURE (Renal and urinary disorders) | 1 (1)
GYNAECOMASTIA (Reproductive system and breast disorders) | 1 (1)
PELVIC PAIN (Reproductive system and breast disorders) | 1 (1)
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 2 (2)
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (2)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
HYPERCAPNIA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 2 (2)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 1 (1)
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 1 (1)
LIPODYSTROPHY ACQUIRED (Skin and subcutaneous tissue disorders) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 1 (1)
BENIGN TUMOUR EXCISION (Surgical and medical procedures) | 1 (1)
DENTAL OPERATION (Surgical and medical procedures) | 1 (1)
HERNIA REPAIR (Surgical and medical procedures) | 1 (1)
INGUINAL HERNIA REPAIR (Surgical and medical procedures) | 1 (1)
LEG AMPUTATION (Surgical and medical procedures) | 1 (2)
PHLEBOTOMY (Surgical and medical procedures) | 1 (1)
PULMONARY VALVE REPLACEMENT (Surgical and medical procedures) | 1 (1)
TOOTH EXTRACTION (Surgical and medical procedures) | 1 (1)
HYPERTENSION (Vascular disorders) | 1 (1)
PERIPHERAL ISCHAEMIA (Vascular disorders) | 1 (1)
PHLEBITIS (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Antiretroviral Combination Therapy Including Raltegravir (N=480)
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 27 (27)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No